CLINICAL TRIAL: NCT05926908
Title: Hospital-Induced Immobility - A Backstage Story of Lack of Chairs, Time, and Assistance
Brief Title: Hospital-Induced Immobility
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jan Christensen, Senior researcher, Head of research, Rigshospitalet, Denmark
Other Study IDs: P-2020-1173
Record Dates: First submitted 2023-06-12; First posted 2023-07-03 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: In-hospital Mobility; Geriatric; Immobilization
Keywords: Mobilisation; Rehabilitation; older adults; inactivity; hospitalisation
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Geriatric ward: Interventions are: Patients' self-reported level of mealtime mobilisation, observations of the patients' mobilisation level and environment at mealtimes, focus group interviews with health care professionals at the wards, survey on mobilisation awareness among the nursing staff, a Mobilisation Initiative, and formal education for all nursing staff
  Interventions: Behavioral: A Mobilisation Initiative; Behavioral: Focus Group Interviews; Behavioral: Formal Education; Behavioral: Self-reported Level of Mobilisation; Behavioral: Observations of Patients and the Environment; Behavioral: Awareness of Mobilisation Survey
- Medical ward: Interventions are: Patients' self-reported level of mealtime mobilisation, observations of the patients' mobilisation level and environment at mealtimes, focus group interviews with health care professionals at the wards, survey on mobilisation awareness among the nursing staff, a Mobilisation Initiative, and formal education for all nursing staff
  Interventions: Behavioral: A Mobilisation Initiative; Behavioral: Focus Group Interviews; Behavioral: Formal Education; Behavioral: Self-reported Level of Mobilisation; Behavioral: Observations of Patients and the Environment; Behavioral: Awareness of Mobilisation Survey

INTERVENTIONS:
Behavioral: A Mobilisation Initiative — The Mobilisation Initiative consists of physiotherapists assisting nursing staff in mobilising patients to sit in a chair for breakfast and lunch. This intervention follows the interventions of focus group interviews, formal education, observations of patients and the environment, and awareness of mobilisation survey
Behavioral: Focus Group Interviews — Focus group interviews using a semi-structured interview guide are conducted with health care professionals at the wards to explore the acceptability and demand for the contents of the Mobilisation Initiative, including the identification of facilitators and barriers to mobilisation
Behavioral: Formal Education — Formal education for all nursing staff employed at the two wards includes information on the consequences of immobilisation, with the purpose of enhancing confidence, competencies, and awareness of mobilisation
Behavioral: Self-reported Level of Mobilisation — Patient's self-reported mealtime mobilisation level reported through interview-based surveys, including structured follow-up questions
Behavioral: Observations of Patients and the Environment — During breakfast and lunch, the mobilisation status of all patients in the wards is observed using an observation checklist
Behavioral: Awareness of Mobilisation Survey — To assess the nursing staff's awareness of and confidence in the mobilisation of the patients, a short survey on mobilisation awareness is distributed to the nursing staff at both wards

SUMMARY:
Inactivity and bedrest during hospitalisation have numerous negative consequences, and it is especially important that older patients are mobile during hospitalisation. In this study the investigators aimed to identify whether the introduction of formal education of clinical staff and a Mobilisation Initiative could increase mobilisation of patients in a geriatric and a medical ward. Furthermore, the investigators wanted to explore patients' and health care staffs' view on facilitators and barriers for mobilisation during hospitalisation

DETAILED DESCRIPTION:
Staying in bed and being inactive during hospitalisation can lead to a range of adverse consequences especially among older adults. The consequences include loss of muscle mass and strength leading to problems with loss of functional independence, risk of re-hospitalisation, and death. Moreover, older adults do not recover as well as younger adults with poor long-term recovery. The lack of in-hospital mobilisation is due to several factors including the hospital culture and organisational factors. Therefore, it is necessary to bring attention to this problem among the hospital staff. The aim of this study is to identify whether the introduction of formal education of clinical staff and a Mobilisation Initiative can increase the number of patients mobilised for breakfast and lunch among patients admitted to geriatric and medical wards. The activities planned in this study is self-reported level of mealtime mobilisation and observations of the patients, focus group interviews and survey on mobilisation awareness among the clinical staff, introduction of formal education and a Mobilisation Initiative. As hypothesized, this will result in an increased awareness of in-hospital mobilisation leading to an increase in the number of patients mobilised at mealtimes. Accordingly, expectations are that this will affect the activity level of the hospitalised patients and reduce adverse consequences leading to an increase in functional independence and reduce the number of readmissions resulting in a socioeconomic benefit.

ELIGIBILITY:
Inclusion Criteria:

* In-hospital patients in the geriatric and medical ward at Copenhagen University Hospital, Rigshospitalet

Exclusion Criteria:

* Patients declared moribund or delirious in the electronical medical journal
* Patients isolated in the hospital room
* Patients requiring interpreter for communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the geriatric and medical wards at Copenhagen University Hospital, Rigshospitalet
Sampling Method: Probability Sample
Enrollment: 596 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in patients mobilised at lunch | One, two, three, four, five, and six months
  Change in percentage of patients mobilised at lunch t0-t1 Change in percentage of patients mobilised at lunch t1-t2 Change in percentage of patients mobilised at lunch t2-t3 Change in percentage of patients mobilised at lunch t3-t4 Change in percentage of patients mobilised at lunch t4-t5 Change in percentage of patients mobilised at lunch t5-t6
Change in patients mobilised at breakfast | One, two, three, four, five, and six months
  Change in percentage of patients mobilised at breakfast t0-t1 Change in percentage of patients mobilised at breakfast t1-t2 Change in percentage of patients mobilised at breakfast t2-t3 Change in percentage of patients mobilised at breakfast t3-t4 Change in percentage of patients mobilised at breakfast t4-t5 Change in percentage of patients mobilised at breakfast t5-t6

SECONDARY OUTCOMES:
Change in chairs present bedside at breakfast | Two, three, four, five, and six months
  Change in percentage of chairs observed placed bedside at breakfast for each patient t1-t2 Change in percentage of chairs observed placed bedside at breakfast for each patient t2-t3 Change in percentage of chairs observed placed bedside at breakfast for each patient t3-t4 Change in percentage of chairs observed placed bedside at breakfast for each patient t4-t5 Change in percentage of chairs observed placed bedside at breakfast for each patient t5-t6
Change in chairs present bedside at lunch | Two, three, four, five, and six months
  Change in percentage of chairs observed placed bedside at lunch for each patient t1-t2 Change in percentage of chairs observed placed bedside at lunch for each patient t2-t3 Change in percentage of chairs observed placed bedside at lunch for each patient t3-t4 Change in percentage of chairs observed placed bedside at lunch for each patient t4-t5 Change in percentage of chairs observed placed bedside at lunch for each patient t5-t6
Self-reported level of mobilisation | One and six months
  Level of patient's mealtime mobilisation level reported through interview-based surveys on a 5-item ordinal scale: independently, with supervision, with the physical help of one person, with the physical help of two persons, or never sit in a chair.
The Mobilisation Initiative | One and six months
  The utilisation of the Mobilisation Initiative recorded as the daily number of patients referred to and mobilised in the Mobilisation Initiative at each ward
Formal Education | Four and five months
  The number of nursing staff attending formal education
Focus Group Interviews | Two months
  Description of facilitators and barriers for mobilising the patients at each ward
Awareness of mobilisation among the nursing staff | Two months and follow up at eight months
  Levels of awareness on mobilisation among the nursing staff at each ward reported through questionnaires including the questions: "Do you feel confident mobilising your patients to sit in a chair at mealtimes?," "To what degree do you feel prepared to do a safe transfer from the bed to a chair with a patient you do not know?," and "How often do you talk to your colleagues about mobilisation?". Questions are answered on 5-item Likert scales: never, less than half of the time, half of the time, more than half of the time, and every time; and to a very low degree, to a low degree, neither/nor, to a high degree, and to a very high degree

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piper KS, Oxfeldt M, Pedersen MM, Christensen J. Hospital-induced immobility - a backstage story of lack of chairs, time, and assistance. BMC Geriatr. 2024 Aug 24;24(1):704. doi: 10.1186/s12877-024-05286-6. PMID 39182057
- See also: Related Info — https://bmcgeriatr.biomedcentral.com/articles/10.1186/s12877-024-05286-6